CLINICAL TRIAL: NCT07245862
Title: Evaluation of a Family-centered Program for Problematic Gaming/Excessive Screen Use in a Child and Adolescent Population Within Social Services in Light of the New Social Services Law
Brief Title: Evaluation of a Family-centered Program for Problematic Gaming/Excessive Screen Use
Acronym: S-FAME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-05262-01
Record Dates: First submitted 2025-09-12; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Adolescent Behavior; Social Media Addiction; Gaming Disorder; Family Relations
MeSH Terms: conditions — Adolescent Behavior; Internet Addiction Disorder

STUDY DESIGN:
Intervention Model Description: This study is a 2-arm, parallel-group randomized controlled trial (RCT). Social services in three municipalities (Lund, Eslöv) have endorsed the project and provided each a letter of intent. Families seeking help for conflicts related to child digital media use will be invited to participate. Eligible families will be randomly assigned to either the intervention group, receiving the S-FAME program, or the control group, receiving standard care. These groups will be matched based on specific preexisting characteristics. Based on power analyses appx 176 participants will be required to detect a small effect size (d = .03), accounting for potential attrition.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): The critical components include psychoeducation, cognitive restructuring, and social and emotional learning. The goals are to help children and parents understand the positive and negative aspects of screen use and to prevent related problems and family conflicts. The intervention consist of 4 group mettings parents and children separate. Max 10 children per group
  Interventions: Behavioral: Family-centered Program for Problematic Gaming/Excessive Screen Use in a child and adolescent population within Social Services
- Control (Active Comparator): This group will recieve treatment as usual. After final follow up this group will be offered an online parental intervention of 3 sessions
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Family-centered Program for Problematic Gaming/Excessive Screen Use in a child and adolescent population within Social Services — The critical components include psychoeducation, cognitive restructuring, and social and emotional learning.his would be the first intervention offering help for both children and their parents. Such an intervention could be beneficial not only to individual families, but also to society at large by reducing societal costs, enhancing family well-being, and addressing health inequalities . the intervention is agroup intervention in 4 sessions with parents in one group and children in one group. The goals are to help children and parents understand the positive and negative aspects of screen use and to prevent related problems and family conflicts. T
  Arms: Intervention
Behavioral: Control — This group will recieve TAU == treat ment as usual depending on the practice at the Social service they belong to
  Arms: Control

SUMMARY:
The Family-Centered Program for Problematic Gaming and Excessive Screen Use (FAME) is a pioneering initiative designed to address the growing challenges of excessive screen use and gaming among children and adolescents, particularly within family dynamics.

DETAILED DESCRIPTION:
The Family-Centered Program for Problematic Gaming and Excessive Screen Use (FAME) is a pioneering initiative designed to address the growing challenges of excessive screen use and gaming among children and adolescents, particularly within family dynamics. With digital media becoming one of the most prevalent leisure activities, excessive use has been linked to adverse outcomes, including depression, sleep disturbances, and family conflicts. Despite these concerns, there are no evaluated family-centered interventions in Sweden that address these issues comprehensively. This randomized controlled trial (RCT) aims to evaluate the effectiveness and feasibility of the S-FAME program, developed in collaboration with social services across two municipalities (Lund, Eslöv). The program integrates psychoeducation, cognitive restructuring, and social-emotional learning, focusing on both children and their families. It acknowledges that problematic screen use often develops within family contexts and aims to improve parenting practices and enhance parent-child relationships. The project aligns with the new Social Services Act, which will come into effect in July 2025, emphasizing easily accessible, preventive, and low-threshold interventions-so-called non-means-tested services. By targeting both individual and family needs, the intervention has the potential to reduce societal costs, enhance family well-being, and address health inequalities. With its innovative and scalable design, S-FAME provides a much-needed framework to tackle one of today's most pressing challenges in youth development- excessive screen use. We are a team of researchers with great experience in research as well as clinical work in the field of adolescence, social work and ANDTS (Alkohol, narkotika, droger, tobak och spel). The project is well established within the School of Social Sciences/Medical Faculty at Lund University, as well as within the innovation and development departments of two social services units. PI Emma Claesdotter-Knutsson (ECK), associate professor and senior consultant in child and adolescent psychiatry at Lund University/Region Skåne with major research areas of gaming, gambling and screens use. ECK has extensive clinical expertise and has played a key role at the Swedish Public Health Agency, contributing to the development of recommendations on child digital media use. PI ECK brings extensive experience and formal training in leading collaborative projects.

ELIGIBILITY:
Inclusion Criteria:

* family conflicts related to screen use
* spaeks and udnerstand swedish

Exclusion Criteria:

* se above

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
FCU | Baseline; Post treatment; 1 month post treatment
  five items measure parent-child warmth, and three items measure parent-child conflicts

SECONDARY OUTCOMES:
SCREENS-Q (adapted) time (19) • PARCA for assessing aspects of parent-child relationship and parenting practices (22) • FCU five items measure parent-child warmth, and three items measure parent-child conflicts (23) | Baseline; Post treatment; 1 month post treatment
  screening form, for valuing children and adolescent´s screen time screening form, for valuing children and adolescent´s screen time screening form, for valuing children and adolescent´s screen time
PARCA | Baseline; Post treatment; 1 month post treatment
  for assessing aspects of parent-child relationship and parenting practices

CONTACTS AND LOCATIONS:
Locations (1):
- Child and Adolescent Psychiatry Clinic, Lund, Sweden